CLINICAL TRIAL: NCT05345782
Title: Laparoscopic Combined Hypo Gastric Neural Plexus Block and Uterosacral Nerve Block for Patients With Chronic Idiopathic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, ASSITANT PROFESSOR, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00006379 ANESTHESIA
Record Dates: First submitted 2022-03-24; First posted 2022-04-26 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Chronic Idiopathic Pain Syndrome
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Hypo gastric Neural Plexus Block (Active Comparator): laparoscopy for diagnosis of the causes of chronic pelvic pain then injecting 5 ml normal saline for hydro dissection of the retroperitoneal space at the level of the sacral promontory then30 ml (14 ml Marcaine +14 ml normal saline+2ml betamethasone) are injected.
  Interventions: Drug: MARCAINE AND BETAMETHAZONE 1
- Laparoscopic Combined Hypo gastric Neural Plexus Block and Uterosacral Nerve Block (Active Comparator): laparoscopy for diagnosis and conventional surgical treatment of the causes of pelvic pain then injecting 5 ml normal saline for hydro dissection of the retroperitoneal space at the level of the promontory followed by 30 ml (14 ml Marcaine +14 ml normal saline+2ml betamethasone) then injecting 5 ml ( 2.5 marcaine+1ml betamethasone +1.5 ml normal saline) 2 cm away from the cervix at the uterosacral ligament on each sides.
  Interventions: Drug: MARCAINE AND BETAMETHAZONE 2

INTERVENTIONS:
Drug: MARCAINE AND BETAMETHAZONE 1 — Laparoscopic Hypo gastric Neural Plexus Block
  Arms: Laparoscopic Hypo gastric Neural Plexus Block
Drug: MARCAINE AND BETAMETHAZONE 2 — Laparoscopic Combined Hypo gastric Neural Plexus Block and Uterosacral Nerve Block
  Arms: Laparoscopic Combined Hypo gastric Neural Plexus Block and Uterosacral Nerve Block

SUMMARY:
Often the etiology of chronic pelvic pain is not clear, as there are many disorders of the reproductive tract, gastrointestinal system, urological organs, musculoskeletal system, and psych neurological system that may be associated with chronic pelvic pain.

An effective treatment for this condition has evaded the medical profession for centuries. Even today only 20-25% patients respond to conservative management.5 When such treatment fails, a diagnostic laparoscopy is performed.1, 3, 6 the cause of the pain is not always obvious as no pathology is seen in 40-60% of the cases.1

DETAILED DESCRIPTION:
This prospective randomized controlled study will be conducted at Eldemerdash hospital. 60 patients will be included with the following criteria:

. Intraoperatively, all patients were monitored by standard monitoring.

All Patients will be assigned randomly by using computerized program to one of the two equal groups. Patients will be (thirty patients per group):

Group A ; thirty patients will do laparoscopy for diagnosis of the causes of chronic pelvic pain then injecting 5 ml normal saline for hydro dissection of the retroperitoneal space at the level of the sacral promontory then30 ml (14 ml Marcaine +14 ml normal saline+2ml betamethasone) are injected.

Group B; thirty patients will do laparoscopy for diagnosis and conventional surgical treatment of the causes of pelvic pain then injecting 5 ml normal saline for hydro dissection of the retroperitoneal space at the level of the promontory followed by 30 ml (14 ml Marcaine +14 ml normal saline+2ml betamethasone) then injecting 5 ml ( 2.5 marcaine+1ml betamethasone +1.5 ml normal saline) 2 cm away from the cervix at the uterosacral ligament on each sides.

Pain score ( visual analogue score) was assessed before surgery (basal) and after completion of laparoscopy 4hr, 12hr, 24hr, 48hr, 1, 4, 8,12, 16,20 and 24 weeks.

Visual analogue scale:

No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10 Duration of pelvic pain relieve after laparoscopy up to 16 weeks,side effects like urinary retention, constipation were recorded after completion of laparoscopy 4hr, 12hr, 24hr, 48hr, 1week, 4weeks, 8 weeks, 12 weeks and 16 weeks.

Urinary retention will be treated by reassuring the patients and catheterization as it usually resolves after 2-3 days, constipation will be treated by reassuring the patients and purgatives as it usually resolves after 2-3 days.

Postoperatively, all patients were transferred to postoperative care unit (PACU) and monitored every 10 min until discharge.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 50 years old.

  * American Society of Anesthesiologists physical status (ASA-PS) I and II Patients.
  * Sex: female.
  * Patients scheduled for elective laparoscopy for diagnosis of the cause of chronic pelvic pain.

Exclusion Criteria:

* • Patient refusal.

  * Patients on chronic pain medications.
  * ASA III or worse clinical condition.
  * Intra-abdominal infection.
  * Allergy to any of the study medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-04-26 (Estimated); Study Completion 2023-04-26 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score | before laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 4 hours after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 12 hours after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 24 hours after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 48 hours after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 1st week after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 4th week after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 8th week after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 12th week after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10
Visual analogue score | 16th week after laparoscopy
  Visual analogue scale:
  No pain Moderate Worst Pain 0 1 2 3 4 5 6 7 8 9 10

SECONDARY OUTCOMES:
constipation(number of patients) | up to 16 weeks postoperatively
urinary retention (number of patients) | up to 16 weeks postoperatively
duration of pain relieve | up to 16 weeks postoperatively
Duration of pelvic pain relieve | up to 16 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: AIN SHAMS UNIVERSITY, Study Chair — asuh
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No